CLINICAL TRIAL: NCT05689684
Title: Arabinoxylan-oligosaccharides (AXOS) As a Medical Food for Adjuvant Approach in the Management of Type-2 Diabetes
Brief Title: Arabinoxylan-oligosaccharides (AXOS) for the Management of Type-2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Carbiotix AB (Industry); Skane University Hospital (Other); Vinnova (Other Government)
Responsible Party: Principal Investigator, LieseLotte Cloetens, Senior Lecturer, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AXOS22; 2022-05204 (Other Grant/Funding Number: Vinnova)
Record Dates: First submitted 2022-12-21; First posted 2023-01-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Type 2
Keywords: AXOS; AG; XOS; metformin; gut microbiome; corn bran extract
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid Product: Aarabinogalactan (AG)+xylan-oligosaccharides (XOS) +AXOS (Active Comparator): Daily 2x 5g Hybrid Product, produced by Carbiotix AB. Hybrid Product is available as powder, which can be easily dissolved in water.
  Interventions: Dietary Supplement: AG+XOS+AXOS
- Placebo (Placebo Comparator): Daily 2x 5g maltodextrin. Maltodextrin is available as powder, which can be easily dissolved in water.
  Interventions: Dietary Supplement: Placebo Maltodextrin

INTERVENTIONS:
Dietary Supplement: AG+XOS+AXOS — 4-month parallel randomized controlled study
  Arms: Hybrid Product: Aarabinogalactan (AG)+xylan-oligosaccharides (XOS) +AXOS
Dietary Supplement: Placebo Maltodextrin — 4-month parallel randomized controlled study
  Arms: Placebo

SUMMARY:
The project aims to achieve significantly improved clinical care for type 2 diabetes. The current standard treatment metformin has low adherence due to its main side effect gut dysbiosis, which also results in more complications and high overall costs. Prebiotics have been suggested as a medical food and might be helpful as adjuvant management in type 2 diabetes and other metabolic diseases. Carbiotix AB has developed, a corn fiber extract containing arabinoxylan-oligosaccharides (AXOS), which have great potential for improving gut health. In this project, it will be investigated whether the intake of a hybrid product containing AXOS together with metformin can significantly improve glucose metabolism and gut health in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (T2D) is a high prevalence and the leading cause of death and disability worldwide. The quality of life is significantly decreased in these patients and the costs for medical care are enormous. T2D patients are often treated with metformin, but adherence to the treatment is relatively poor, with gut dysbiosis as a major cause. Gut dysbiosis has not been addressed in the clinical setting although numerous studies support its role in disease development. There is an urgent need to improve existing treatments with metformin to improve adherence to drug therapy and the management of the disease. Prebiotics are dietary fibers that stimulate the growth and activity of beneficial gut microbiota. Prebiotics has been suggested as a medical food and might be very useful as an effective adjuvant approach in the management of T2D and other metabolic diseases. Carbiotix AB, a biotech company based in Lund, has developed a corn fiber extract containing arabinoxylan-oligosaccharides (AXOS), which have great potential for improving gut health.

In this project, a clinical trial will be performed to investigate whether the corn fiber extract can significantly increase metformin adherence with improved gut health and glucose metabolism in patients with T2D. To maximize the potential efficacy of the intervention, a "Hybrid Product" containing arabinogalactan (AG), xylan-oligosaccharides (XOS), and AXOS will be used, building on the XOS and AXOS naturally present in the corn fiber extract.

One hundred subjects with T2D and treated with metformin will be recruited for this blind parallel randomized controlled intervention study. After a screening visit, the subjects will be randomized to test the Hybrid Product or placebo (maltodextrin) group. The duration of the intervention is 4 months, and the study subjects will be asked to consume the Hybrid Product or placebo daily (2x 5g). At the start, of week 8 and week 16, the study subjects will visit the study center for the measurement of body weight, waist circumference, and blood pressure. At these 3 visits, fasting blood samples are taken for analysis of glucose and insulin metabolism, blood lipids, and inflammation markers. Fecal samples are also collected to investigate the effect of the Hybrid Product on microbiota composition. At regular times during the study, the subjects must do a 7-point blood glucose monitoring and fill in questionnaires about gastrointestinal symptoms. During the whole study period, all subjects are contacted regularly to follow up on their health status.

If the Hybrid Product shows the strong potential to improve adherence to metformin treatment, this will lead to improving diabetes care with reduced economic consequences. The promotion of a healthy gut by consumption of soluble fibers also helps to support immune function, blood sugar regulation, increased nutrient uptake (e.g. vitamin B12), and better body weight control. These health benefits will undoubtedly result in better well-being in private and working life and thus in a significantly improved quality of life for patients with T2D. Furthermore, effective treatment of T2D will also reduce the prevalence of cardiovascular risk factors, which are key targets in the current public health debate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with T2D and taking metformin as treatment for at least 6 months
* Age 50-80 years, at the time of signing the informed consent
* BMI 25-40 kg/m2
* Stable body weight (less than 5% difference during the last 3 months)
* Willing and able to give written informed consent for participating the study
* Willing to comply with all study procedures

Exclusion Criteria:

* Hba1c > 60 mmol/L
* fP-triglycerides > 4 mmol/ L - can be included if stabilized by medication
* fP total cholesterol >8 mmol/L - can be included if stabilized by medication
* high blood pressure >160/90 mmHg - can be included if stabilized by medication
* intake of antibiotics within 4 weeks prior to the start of the study
* regular intake of probiotics and/or prebiotics within 4 weeks prior to the start of the study
* alcohol abuse > 40g/d
* chronical disease (liver, kidney)
* gastrointestinal disease (ulcerative colitis, Crohn's disease, irritable bowel syndrome)
* heart disease (within the last 12 months)
* treatment with corticosteroids of significant degree
* psychological disease of significant degree
* cancer of significant degree
* gastric-bypass operation
* operation planned during the study period
* known gluten intolerance, lactose intolerance, milk protein allergy
* other food allergy
* special diet (e.g. vegetarian, vegan, LCHF, 5-2)
* non-Swedish speaking and reading
* investigator considers the subject unlikely to comply with the study procedures, restrictions, and requirements

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
change in levels of postprandial blood glucose | 0, 2months and 4months
  Postprandial blood glucose will be analysed at the university hospital according to standard analytical procedures

SECONDARY OUTCOMES:
gastrointestinal symptoms (bloating, abdominal pain, diarrhea, constipation) | 0, 1months, 2months, 3months, 4months
  Gastrointestinal symptoms will be measured using a questionnaire with a scale 0-5
composition and activity of the gut microbiota (genus and species) | 0, 2months and 4months
  Fecal samples will be analysed to measure microbiota composition using high-throughput next-generation sequencing of 16S rRNA amplicons and quantitative PCR
levels of fasting blood glucose | 0, 2months and 4months
  Blood samples will be taken and analysed for glucose at the university hospital according to standard analytical procedures
level of Hba1c | 0, 2months and 4months
  Blood samples will be taken and analysed for Hba1c at the university hospital according to standard analytical procedures
blood lipid profile | 0, 2months and 4months
  Blood samples will be taken and analysed for total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides at the university hospital according to standard analytical procedures
immune functions | 0, 2months and 4months
  Blood samples will be taken and analysed for CRP at the university hospital according to standard analytical procedures
uptake of vitamin B12 and vitamin D | 0, 2months and 4months
  Blood samples will be taken and analysed for vitamin B12 and vitamin D at the university hospital according to standard analytical procedures
systolic and diastolic blood pressure | 0, 2months and 4months
  Systolic and diastolic blood pressure will be measured twice in sitting position using automatic devices
body weight | 0, 2months and 4months
  Body weight will be measured in kg to the nearest 0,1 kg using a digital scale

CONTACTS AND LOCATIONS:
Overall Officials: Lieselotte Cloetens, Principal Investigator — Lund University
Locations (1):
- Biomedical Nutrition, Lund University and Department of Endocrinology , Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boll EV, Ekstrom LM, Courtin CM, Delcour JA, Nilsson AC, Bjorck IM, Ostman EM. Effects of wheat bran extract rich in arabinoxylan oligosaccharides and resistant starch on overnight glucose tolerance and markers of gut fermentation in healthy young adults. Eur J Nutr. 2016 Jun;55(4):1661-70. doi: 10.1007/s00394-015-0985-z. Epub 2015 Jul 14. PMID 26169871
- [Background] Cloetens L, Broekaert WF, Delaedt Y, Ollevier F, Courtin CM, Delcour JA, Rutgeerts P, Verbeke K. Tolerance of arabinoxylan-oligosaccharides and their prebiotic activity in healthy subjects: a randomised, placebo-controlled cross-over study. Br J Nutr. 2010 Mar;103(5):703-13. doi: 10.1017/S0007114509992248. Epub 2009 Dec 10. PMID 20003568
- [Background] Gibson GR, Hutkins R, Sanders ME, Prescott SL, Reimer RA, Salminen SJ, Scott K, Stanton C, Swanson KS, Cani PD, Verbeke K, Reid G. Expert consensus document: The International Scientific Association for Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of prebiotics. Nat Rev Gastroenterol Hepatol. 2017 Aug;14(8):491-502. doi: 10.1038/nrgastro.2017.75. Epub 2017 Jun 14. PMID 28611480
- [Background] McGovern A, Tippu Z, Hinton W, Munro N, Whyte M, de Lusignan S. Comparison of medication adherence and persistence in type 2 diabetes: A systematic review and meta-analysis. Diabetes Obes Metab. 2018 Apr;20(4):1040-1043. doi: 10.1111/dom.13160. Epub 2017 Dec 12. PMID 29135080
- [Background] Uusitupa M, Khan TA, Viguiliouk E, Kahleova H, Rivellese AA, Hermansen K, Pfeiffer A, Thanopoulou A, Salas-Salvado J, Schwab U, Sievenpiper JL. Prevention of Type 2 Diabetes by Lifestyle Changes: A Systematic Review and Meta-Analysis. Nutrients. 2019 Nov 1;11(11):2611. doi: 10.3390/nu11112611. PMID 31683759